CLINICAL TRIAL: NCT07306390
Title: Distribution and Analysis of Metastatic Lymph Nodes in Colorectal Cancer Patients (DIAMOND)
Acronym: DIAMOND
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); Shanxi Province Cancer Hospital (Other); The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, HAI ZENG ZHAGN, Medical Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: 25/631-5577
Record Dates: First submitted 2025-11-25; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colorectal Cancer; Lymph Node Metastasis; Spatial Distribution
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Cancer Patients

SUMMARY:
The goal of this observational study is to learn about the spatial distribution and significance of metastatic lymph nodes in colorectal cancer patients. The main question it aims to answer is:

* What is the spatial distribution pattern of metastatic lymph nodes in patients with colorectal cancer?
* Can the spatial distribution pattern of metastatic lymph nodes in patients with colorectal cancer guide clinical practice? Participants should undergo regular follow-up examinations for at least 5 years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* Pathologically confirmed adenocarcinoma of the colon or rectum
* Underwent radical resection for colorectal cancer with a D3 lymphadenectomy and lymph nodes were submitted for pathological examination according to standardized station-based and distance-based protocol
* No distant metastasis or distant metastasis within 6 months after surgery
* No history of other malignant tumors or severe systemic diseases
* No immune diseases or inflammatory bowel diseases
* Non-emergency surgery
* With complete clinicopathological and follow-up data

Exclusion Criteria:

* Pathologically confirmed benign tumors or non-adenocarcinoma malignancies
* Underwent local excision or palliative resection
* Regional lymph nodes were not dissected or submitted for pathological examination according to the unified station-based or distance-based protocol
* With distant metastasis or distant metastasis within 6 months after surgery
* Dual or multiple primary colorectal cancers or concurrent other malignant tumors
* Had a previous diagnosis of immune diseases or inflammatory bowel disease such as ulcerative colitis or Crohn's disease
* Underwent emergency surgery
* Had incomplete clinicopathological or follow-up data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients who undergo radical resection in the National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, China-Japan Friendship Hospital, Shanxi Cancer Hospital, and The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital between December 2025 and December 2027.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The spatial distribution of metastatic lymph nodes | From enrollment to 14 days after surgery (at the completion of postoperative pathological examination)

SECONDARY OUTCOMES:
Disease-free survival | From date of surgery until the date of first documented local recurrence, distant metastasis, or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival | From date of surgery until the date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Haizeng Zhang, Doctorate, Study Chair — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The Institutional Review Board or Ethics Committee may restrict the scope of all individual participant data sharing.